CLINICAL TRIAL: NCT03764397
Title: Development and Piloting of a Prehabilitation Behavioural Change and Physical Activity Intervention for Fibromyalgia Syndrome
Brief Title: Prehabilitation for Being Active. A Feasibility Study in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Fernando Estévez-López, PhD, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/0079
Record Dates: First submitted 2018-11-27; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Fibromyalgia
Keywords: Lifestyle; Education; Self-management; Physical Activity; Proof-of-concept study
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation group (Experimental): A 4-week prehabilitation educational programme (i.e., a behavioral change intervention) and to pilot that prehabilitation in combination with a 6-week gentle self-paced walking programme (with weekly telephone support) in people with FM.
  Interventions: Behavioral: Prehabilitation for behavioural change

INTERVENTIONS:
Behavioral: Prehabilitation for behavioural change — The 4-week prehabilitation educational programme will consist of a meeting for one session (approximately 1 - 1.5 hours) per week. This behavioural change programme will involve a mixture of interactive and didactic sessions, facilitated by a physiotherapist, psychologists, and other health professionals. The purpose of the initial prehabilitation programme is to gain participant 'buy-in' to the programme, to assist participants engage with exercise, to help participants overcome barriers to exercise and improve self-efficacy for exercise. The prehabilitation phase will also enable participants to understand why and how to perform gentle self-paced exercise. After the prehabilitation programme, participants will be advised to engage in a 6-week gentle self-paced walking programme; i.e., a simple pedometer-driven walking programme with weekly telephone support.

SUMMARY:
Twelve people with FM will be recruited from the FM patient support groups. The investigators will develop and test a 4-week prehabilitation educational programme (i.e., a behavioural change intervention) consisting of meeting once per week (each approximately 1 - 1.5 hours). These dynamic and interactive meetings will focus on education and skills training in: exercise, activity cycling, pacing, causes of symptoms in FM (pain, fatigue, sleep dysfunction) and their management.

Participants will be taught to set specific, measurable, achievable, realistic and timed goals (SMART principle) that are valuable or meaningful to them. To do so, the participants will identify a 'committed action' plan. The principles of cognitive behavioural therapy will be used to address maladaptive thoughts (e.g., catastrophizing and fear avoidance) and to manage stress (e.g., skills of relaxation). Participants will learn how to use of pedometers to monitor physical activity.

After the 4-week prehabilitation educational programme, the participants will be encouraged to engage in a 6-week gentle self-paced walking programme (with weekly telephone support).

The 6-week walking programme will consist of a simple pedometer-driven intervention.

Furthermore, the research team will telephone each participant at a prearranged time each week to discuss progress, to document mean daily step count and to discuss a new physical activity target (step count) for the subsequent week. Participants will record daily step counts (pedometer-derived) in a walking dairy which will be used as raw data and mean steps per day calculated. Where a participant declines telephone support, an alternative weekly email or text/WhatsApp messages will be offered instead, where the same information will be given and requested.

Before (baseline measurements) and right after the completion of the 4-week prehabilitation educational programme as well as the 6-week gentle self-paced walking programme the same measurements will be taken. By doing so, the investigators will evaluate short and mid-term changes promoted by the prehabilitation programme. The participants will fill out the following questionnaires: the Revised FM Impact Questionnaire, Pain Catastrophizing Scale, Multidimensional Fatigue Inventory, Short-Form 36-item Health Survey, International Physical Activity Questionnaire, Sedentary Behaviour Questionnaire, Exercise Self Efficacy Questionnaire, Pittsburgh Sleep Quality Index questionnaire, and the modified 2011 preliminary FM criteria questionnaire.

Right after the completion of the prehabiliation intervention, all the participants will fill out the treatment acceptability and credibility questionnaire. Right after the completion of the walking programme, participants will be interviewed (semistructured face-to-face exit interview lasting about 30-45 minutes) to explore their experiences of the study including barriers to participation.

The main outcome of the study will be acceptability and credibility of the prehabilitation intervention (treatment acceptability and credibility questionnaire. Additionally, the success of the prehabilitation programme will be based on (i) number of sessions attended (>80%), (ii) number of drop outs (<15%) and reasons for early withdrawal, (iii) number of screening questionnaires completed and returned (>80%).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with FM by a medical practitioner, which will be confirmed by the research team -i.e., the modified 2011 preliminary FM criteria questionnaire (Appendix 14) by satisfying 'widespread pain index' (WPI) and 'symptom severity scale' (SS) as follows, either WPI ≥7 and the SS ≥5, or the WPI is 3-6 and the SS ≥9.

Exclusion Criteria:

* Younger than 16 years old.
* Not able to communicate in English.
* Mobilise dependently/aided.
* Have any medical condition that would make exercise participation unsafe (for example; heart disease, stroke, respiratory disease, severe mobility problems, severe arthritis or inflammatory joint disease).
* Are involved in ongoing litigation involving FM.
* Are currently under active treatment by a physiotherapist or involved in any other research studies.
* Are pregnant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Acceptability and credibility of the prehabilitation intervention | Time point(s): once, right after the education programme. Time frame: An average of the past 4 weeks
  The treatment acceptability and credibility questionnaire
Number of sessions attended | Time point(s): once, right after the education programme. Time frame: The past 4 weeks
  Percentage of participants attending to more than 80% of the education sessions
Number of drop outs and reasons for early withdrawal | Time point(s): once, right after the education programme. Time frame: The 4 past weeks
  Percentage of participants that do complete the study
Number of questionnaires completed and returned | Time point(s): once, right after the education programme. Time frame: The 4 past weeks
  Percentage of participants that complete and return, at least, 80% of the questionnaires

SECONDARY OUTCOMES:
Severity of fibromyalgia (also know as, impact of fibromyalgia) | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: The past week
  the Revised FM Impact Questionnaire
Pain intensity | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: The past week
  0-10 NRS
Pain catastrophizing | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: "in general", an average of the past 4 weeks.
  Pain catastrophizing is the tendency to describe a pain experience in more exaggerated terms than the average person, to ruminate on it more (e.g., "I kept thinking 'this is terrible'"), and/or to feel more helpless about the experience ("I thought it was never going to get better"). Pain catastrophizing will be measured by means of the Pain Catastrophizing Scale is a 13-item questionnaire in which patients are asked to reflect on past painful experiences and indicate their thoughts or feelings about pain, on a 5-point scale. For this study, the total score (range 0-52) was used, where higher scores represent a more negative appraisal of pain.
Fatigue | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: The past week
  the Multidimensional Fatigue Inventory
health related quality of life | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: "in general", an average of the past 4 weeks.
  the Short-Form Health Survey
physical activity | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: the past 7 days
  the International Physical Activity Questionnaire
Sedentary Behaviour | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: the past week
  Sedentary Behaviour Questionnaire
exercise self-efficacy | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: "in general", an average of the past 4 weeks.
  the Exercise Self Efficacy Questionnaire
sleep quality | Time point(s): 3 (baseline, 4th and 10th weeks). Time frame: "in general", an average of the past 4 weeks.
  the Pittsburgh Sleep Quality Index questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Hughes, PhD, Principal Investigator — Ulster University
Locations (1):
- The VINE center, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Derived] Courel-Ibanez J, Estevez-Lopez F, Hughes C, Adams N, Fullen BM, Davison G, Montgomery A, Cramp F, Maestre C, Martin D, McVeigh JG. Proof of concept of prehabilitation: a combination of education and behavioural change, to promote physical activity in people with fibromyalgia. BMJ Open. 2023 Jul 14;13(7):e070609. doi: 10.1136/bmjopen-2022-070609. PMID 37451740